CLINICAL TRIAL: NCT00836732
Title: MESenchymal Stem Cells: Alterations in GEnome
Acronym: MESSAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BRD 08/9-S
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Pened Chest Surgery for Programmes Coronary Bypass
Keywords: celle therapy; cell culture; mesenchymal stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: harvest of a small bone marrow sample — harvest of a small bone marrow sample during open chest surgery

SUMMARY:
The aim is to study small genetic alterations induced by cell culture in human mesenchymal stem cells in GMP condition.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 old
* age < 75 old
* opened chest surgery for programmed coronary bypass

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Presence of small genetic alteration in mesenchymal stem cells | one month

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lemarchand, MD, Principal Investigator — Nantes UH - institut du thorax
Locations (1):
- nantes University Hospital, Nantes, Nantes, France